CLINICAL TRIAL: NCT02497118
Title: Clinical Study of Recombinant Human Endostatin Combined With NP Chemotherapy in the Treatment of Stage ⅢA Non Small Cell Lung Cancer
Brief Title: Recombinant Human Endostatin Combined With NP in Neoadjuvant Chemotherapy of Stage ⅢA NSCLC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMUCIH-ENDU-S001
Record Dates: First submitted 2015-07-05; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2014-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: lung cancer Anti angiogenesis therapy survival
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Endostatins; endostar protein; Vinorelbine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endostatin plus NP (Experimental): drug:Endostatins Intravenous drip， 7.5mg/m^2, d1-14 drug:vinorelbine Intravenous drip 25mg/m^2,IV, d1, d8; drug:Cisplatin，75mg/m^2 Intravenous drip,divide into d1-3 for 2 cycles
  Interventions: Drug: Endostatin; Drug: Vinorelbine; Drug: Cisplatin
- NP neoadjuvant chemotherapy (Active Comparator): drug:vinorelbine Intravenous drip 25mg/m^2,IV, d1, d8; drug:Cisplatin，75mg/m^2 Intravenous drip,divide into d1-3 for 2 cycles
  Interventions: Drug: Vinorelbine; Drug: Cisplatin

INTERVENTIONS:
Drug: Endostatin — Endostatin,7.5mg/m^2,intravenous, d1-14;
  Other Names: Endostar
  Arms: Endostatin plus NP
Drug: Vinorelbine — vinorelbine,25mg/m^2,intravenous, d1, d8;
Drug: Cisplatin — Cisplatin，75mg/m^2 intravenous,divide into d1-3

SUMMARY:
This study mainly to observe the anti angiogenic drugs Endostatin (Endostar) combined with vinorelbine and Cisplatin (NP) as neoadjuvant therapy in patients with non small cell lung cancer clinical efficiency and safety. Through anti angiogenesis therapy combined with neoadjuvant chemotherapy improve the treatment of neoadjuvant therapy in tumor response rate and the rate of resection, At the same time, the study before and after the anti angiogenesis therapy in patients with peripheral blood circulation endothelial cells(CECs), levels of Endothelial progenitor cells（EPC）, micro vascular density（MVD） and vascular endothelial growth factor(VEGF) expression level, to understanding the correlation between the clinical efficacy of anti angiogenesis therapy combined with chemotherapy and the change of all these markers. In order to find the reference basis for the prediction of the effect of curative effect. The changes of blood volume, blood flow and vascular permeability of the lung cancer before and after treatment with CT perfusion imaging are studied.

ELIGIBILITY:
Inclusion Criteria:

* The pathology proved to be non small cell lung cancer (must be histologically).
* At present, the patients with ⅢA stage (N2) were evaluated by the assistant examination;
* The patients were evaluated by imaging, laboratory examination and other examination;
* Without chemotherapy or anti angiogenic therapy;
* There can be measured lesions
* Informed consent.

Exclusion Criteria:

* Pregnant, lactating women, or patients with fertility but did not take contraceptive measures.
* Severe infection.
* Severe heart disease.Neuropsychiatric disorders, which is not easy to control.
* Severe diabetes.
* There is obvious bleeding tendency.
* The 5 years history of other tumors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Tumor Regression Rate | 3 months
  Target lesion size reduction ratio

SECONDARY OUTCOMES:
Disease free survival is defined as the time from randomization to disease recurrence or death which comes first. | 5 years
Overall Survival | 5 years
  the time from randomization to death.
Clinical Benefit Rate | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Zhao X, Su Y, You J, Gong L, Zhang Z, Wang M, Zhao Z, Zhang Z, Li X, Wang C. Combining antiangiogenic therapy with neoadjuvant chemotherapy increases treatment efficacy in stage IIIA (N2) non-small cell lung cancer without increasing adverse effects. Oncotarget. 2016 Sep 20;7(38):62619-62626. doi: 10.18632/oncotarget.11547. PMID 27566586